CLINICAL TRIAL: NCT06724666
Title: Transdiagnostic Internet-delivered Intervention for Adolescents With Anxiety and Depression
Acronym: NEURO4C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Costina-Ruxandra Poetar, Assistant professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNRR-III-C9-2022-I8-CF278
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders; Depressive Disorder; Social Anxiety Disorder; Major Depressive Disorder; Dysthymia; Generalized Anxiety Disorder
Keywords: Internet-delivered intervention; transdiagnostic; adolescents; internalizing; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Phobia, Social; Depressive Disorder, Major; Dysthymic Disorder; Generalized Anxiety Disorder; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Internet-delivered intervention (Experimental): The intervention consists of 8 modules delivered over 8 weeks. It is based on Rational Emotive Behavioral Therapy (REBT).
  Interventions: Behavioral: Transdiagnostic Internet-delivered intervention
- Control group (No Intervention): Participants in the control group are a delayed intervention group (waiting list control). They will access the intervention after 8 weeks.

INTERVENTIONS:
Behavioral: Transdiagnostic Internet-delivered intervention — The intervention consists of 8 modules based on Rational emotive therapy, delivered via 8 weeks.
  Arms: Transdiagnostic Internet-delivered intervention

SUMMARY:
The goal of this clinical trial is to test the efficacy of a transdiagnostic Internet-delivered interventions for Romanian adolescents with anxiety and/ or depression. The main questions it aims to answer are:

* What is the clinical efficacy of the Internet-delivered intervention?
* How accurate is the prediction model in predicting who will respond to treatment? Participants will undergo non-invasive fMRI to measure variability in brain signal as a proxy of the neural systems' adaptability before receiving the intervention, then they will be allocated either to the Internet-delivered intervention or control group.

DETAILED DESCRIPTION:
To the best of investigators' knowledge, this is the first clinical trial conducted with adolescents diagnosed with anxiety/and or depressive disorders that tests the accuracy of a prediction model based on fMRI to investigate participants' response to a transdiagnostic Internet-delivered intervention.

ELIGIBILITY:
Inclusion Criteria:

* elevated symptoms of anxiety or depression/ internalizing problems (T score> 60) at intake (based on Youth self-report completed by adolescents)
* primary diagnosis of an anxiety/depressive disorder based on DSM-5 criteria according to ADIS-5-C/P interview
* age 13-17
* able to read and understand Romanian language
* Currently unmedicated or on stable and adequate doses of medication for at least 6 weeks before treatment onset
* Internet access

Exclusion Criteria:

* severe mental disorder (psychosis, severe depression, bipolar disorder, based on clinical interview)
* any condition that interferes with the protocol implementation (e.g., physical illness or sensory impairment that interferes with behavioral tasks such as exposure, behavioral activation, unavailable for the next 3 months),
* active suicidal ideation (assessed by child psychiatrist during clinical interview) in the last month
* currently following CBT/ psychotherapy for anxiety/depression, in the last 6 months
* fMRI incompatible (based on safety questionnaire)
* Being diagnosed with an intellectual disability, pervasive developmental disorder, an alcohol and/or substance dependence disorder, reading disabilities (based on clinical interview).
* Current treatment with benzodiazepines

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Internalizing problems | baseline, after 8 weeks of intervention, 6 months follow-up
  Change from baseline in internalizing problems. Revised Children's Anxiety and Depression Scale (RCADS) completed by adolescents.

SECONDARY OUTCOMES:
Clinical diagnosis | administered pre-baseline, post-baseline (after 8 week waitlist period), after 8 weeks of intervention
  Change in DSM-5 Anxiety and Depressive Disorder Diagnoses in Accordance with Anxiety Disorders Interview Schedule for the DSM-5, Child and Parent Versions (ADIS-5-C/P) Clinical Diagnosis
Global functioning | baseline, after 8 weeks of intervention, 6 months follow-up
  Children's Global Assessment Scale (C-GAS)
Severity | baseline, after 8 weeks of intervention, 6 months follow-up
  Clinical Global Impression Scale - Severity
Improvement | after 8 weeks of intervention, 6 months follow-up
  Clinical Global Impression Scale - Improvement
Comorbid problems | baseline, after 8 weeks of intervention, 6 month follow-up
  Subscales of the Revised Children's Anxiety and Depression Scale (RCADS) completed by adolescents
Life satisfaction | baseline, after 8 weeks of intervention, 6 months follow-up
  SWLS-C: Satisfaction with Life Scale for Children
Satisfaction with the Internet-delivered intervention | after 8 weeks of intervention
  Client Satisfaction Questionnaire (CSQ-8)
Working alliance | after 8 weeks of intervention
  Working alliance scale for Internet interventions
Automatic thoughts | baseline, after 8 weeks of intervention, 6 month follow-up
  Automatic thoughts questionnaire
Credibility and expectations | week 2
  Credibility and expectations questionnaire
Credibility and expectations based on primary outcome measure | baseline
  Credibility and expectations based on primary outcome scale
Anxiety and depressive symptoms | baseline, at each 2 weeks during treatment duration, after 8 weeks of intervention, 6 months follow-up
  PHQ4
Avoidance | baseline, after 8 weeks of intervention, 6 month follow-up
  CAMS
Parental distress | baseline
  DASS-21
Adolescent anxiety and depressive symptoms as reported by parents | baseline, after 8 weeks of intervention, 6 month follow-up
  RCADS-47 parent report
Parental accommodations | baseline
  Family accommodation scale - parent report

CONTACTS AND LOCATIONS:
Overall Officials: Costina Poetar, PhD, Study Chair — Babeș-Bolyai University
Locations (2):
- Romania (2):
  - Babes-Bolyai University, Cluj-Napoca
  - Babeș-Bolyai University, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be will be shared after the publication of the results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Supporting information will be shared after the publication of the results.
Access Criteria: Supporting information will be publicly shared in OSF.